CLINICAL TRIAL: NCT01579539
Title: The Effect of Intravenous Glucocorticoids on the Tearfilm in Eyes With Thyroid-associated Ophthalmopathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Ass. Prof. PD. Dr., Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPHT-120312
Record Dates: First submitted 2012-04-13; First posted 2012-04-18 (Estimated); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Thyroid-associated Ophthalmopathy; Dry Eye Syndrome
Keywords: Methylprednisolone; Dry Eye Syndrome; Tear Film; Thyroid-associated ophthalmopathy
MeSH Terms: conditions — Graves Ophthalmopathy; Dry Eye Syndromes | interventions — Methylprednisolone; Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients (Experimental): Patients with moderate to severe thyroid-associated ophthalmopathy
  Interventions: Drug: Methylprednisolone; Drug: Esomeprazole

INTERVENTIONS:
Drug: Methylprednisolone — 500mg i.v. infusion once a week for 6 weeks followed by 250mg i.v. infusion once a week for 6 weeks
Drug: Esomeprazole — 40mg i.v. infusion once a week for 12 weeks

SUMMARY:
Thyroid-associated ophthalmopathy (TAO), also called Graves' ophthalmopathy or thyroid eye disease, is a common orbital disease in adults. Patients with TAO, especially in its active phase, often complain about symptoms of ocular surface discomfort, including excess tearing, gritty sensation, increased sensitivity to light and foreign-body sensation, which are similar to inflammatory ocular surface disorders such as dry-eye syndrome (DES). Incomplete blink, increased proptosis and greater palpebral fissure width in TAO accelerates tear evaporation, which increases the tear fluid's osmolarity, and results in ocular surface damage. The administration of intravenous glucocorticoids can be an effective treatment for TAO.

The rationale of the present study is to assess the effect of intravenously administered glucocorticoids on the signs of DES in patients with TAO with new methods such as measurement of tear film thickness, tear film osmolarity and scattering of the tear film and well established methods for assessment of the severity of DES. Additionally, impression cytology and determination of tear cytokines/chemokines will be performed to obtain information about inflammatory processes on the ocular surface.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged over 18 years
* Active thyroid associated ophthalmopathy with clinical activity score (CAS) of each eye more than 3 or recently experienced worsening of proptosis, lid retraction, or ocular motility disturbance.
* Normal ophthalmic findings except symptoms associated with TAO
* Scheduled for treatment with systemic glucocorticoids according to the kahaly-scheme

Exclusion Criteria:

* Chronic inactive TAO
* Previous treatment with oral or intravenous glucocorticoids 3 months preceding the study
* Participation in a clinical trial in the 3 weeks before the screening visit
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Presence or history of a severe medical condition that will interfere with the study aim as judged by the clinical investigator
* Wearing of contact lenses
* Intake of dietary supplements in the 3 months preceding the study
* Topical treatment with any ophthalmic drug in the 4 weeks preceding the study except topical lubricants
* Ocular infection
* Ocular surgery in the 3 months preceding the study
* Sjögren's syndrome
* Stevens-Johnson syndrome
* Pregnancy, planned pregnancy or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-06-27 (Actual); Primary Completion 2017-05-18 (Actual); Study Completion 2017-05-18 (Actual)

PRIMARY OUTCOMES:
Tear film thickness as measured with OCT | 13 weeks
  Measurements of tear film thickness with OCT will be performed 7 or less days before start of treatment, 6 weeks after start of treatment and 12 weeks after start of treatment

SECONDARY OUTCOMES:
Break up time (BUT) | 13 weeks
Visual acuity | 13 weeks
Tear film osmolarity | 13 weeks
Degree of exophthalmia | 13 weeks
  Hertel exophthalmometry
Palpebral fissure width | 13 weeks
OSI (Objective Scattering Index) | 13 weeks
Tear cytokines/chemokines | 13 weeks
Impression cytology | 13 weeks
Staining of the cornea with fluorescein | 13 weeks
Schirmer I test | 13 weeks
Subjective symptoms of dry eye syndrome | 13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Garhoefer, MD, Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria